CLINICAL TRIAL: NCT04252391
Title: A Randomized Controlled Crossover Study to Determine the Effectiveness of Peri-Neural Electrical Dry Needling (PNED) vs. Standard Care for the Treatment of Patients With Migraine Headaches
Brief Title: Peri-neural Electrical Dry Needling Migraine Treatment Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wheaton Franciscan Healthcare (Other)
Responsible Party: Principal Investigator, Joseph Tepp, Principal Investigator, Wheaton Franciscan Healthcare
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: WheatonFH
Record Dates: First submitted 2020-01-29; First posted 2020-02-05 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Randomized controlled cross-over study
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be masked to which treatment arm they are in. The outcome assessor will be masked to which treatment arm the participant was in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (Active Comparator): Standard care will consist of standard physical therapy care which may include the following: cervical or thoracic manipulation or mobilization, muscle stretching, muscle strengthening, dry needling with or without electrical trigger point dry needling, soft tissue release and prescribed therapeutic exercises .
  Interventions: Procedure: Standard Care
- standard care with perineural electrical dry needling. (Active Comparator): This arm will consist of standard care with perineural electrical dry needling, using a high frequency stimulation placed near the nerve, differing from addressing muscular trigger points. For example, a dry needle placed in the semispinalis capitus muscle along the greater occipital nerve pathway, stimulated at 80 Hz.
  Interventions: Procedure: Perineural electrical dry needling

INTERVENTIONS:
Procedure: Perineural electrical dry needling — Standard care plus use of perineural electrical dry needling involving use of a monofilament needle of 15 or 30 mm length, 0.25 mm diameter will be placed utilizing the therapist's dominant hand following palpation of correct needle location. An electrical stimulation unit will be used to conduct an electrical impulse. The unit used will be an ES-130 by ITO (Japan) using a DC 9V battery producing an asymmetrical biphasic waveform. The unit has 6 available leads with alligator clamps, connecting to needle shafts. Parameters of PNED will include intensity set at a strong yet comfortable setting according to patient feedback. Treatment duration will be 15 minutes. Treatment frequency will be set to Medium at level 8 (80 Hz). Parameters will be set to elicit a sensory response.
  Arms: standard care with perineural electrical dry needling.
Procedure: Standard Care — cervical or thoracic manipulation or mobilization, muscle stretching, muscle strengthening, electrical trigger point dry needling , soft tissue release and prescribed therapeutic exercises .
  Arms: Standard care

SUMMARY:
This study seeks to determine the effectiveness of a specific treatment protocol using dry needling with perineural electrical stimulation in comparison to standard treatment in physical therapy for patients with migraine headaches. This will be a randomized cross-over study in which participants will be in the first arm of the study, have a washout period, then cross over to the other arm of the study.

DETAILED DESCRIPTION:
From current understanding of migraine pathophysiology, the investigators know that it involves excitability of the trigeminovascular system. Intercranial vasculature containing nociceptor innervation consists of unmyelinated (c-fibers) and thinly myelinated (a-delta fibers ) axons which hold vasoactive neuropeptides including substance P and (CGRP) calcitonin gene related peptide. When a migraine occurs, there is a cortical spreading depolarization, which on a molecular level involves a release of ATP, glutamate, potassium, hydrogen ions, glia or vascular cells, and CGRP and nitric oxide by activated perivascular nerves. These substances, including CGRP diffuse to come in contact with nociceptors causing neurogenic inflammation (vasodilation), thus propagating a headache.

Electrical perineural dry needling causes the release of substance-P and CGRG predominantly from non-neural structures, facilitating a negative feedback loop to neural and neuroactive components of the target tissue. This causes a lowering of the levels of CGRP which in turn decreases the inflammatory component thought to play a role in migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 to 100 years old
* Acute or chronic manifestation of migraine headaches or prior diagnosis of migraine headache.
* Numeric pain rating of 3/10 (where 0= no pain and 10= worst pain)

Exclusion Criteria:

* History of epilepsy
* Needle-phobia
* Unstable psychological status
* Compromised immune system
* Metallic allergy
* Having not eaten within the past 3 hours
* Inability to lie in prone, or side-lying
* Pregnant or trying to become pregnant
* Inability to consent or understand English.
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Change in numeric pain rating scale | 1-6 days
  Self reported pain intensity immediately before and after treatment using a numeric pain rating scale from 0 to 10 (0 = no pain and 10 = the worst pain).
  Participants will be assessed 2 days per week with a minimum of 1 day between treatment days.
Change in Neck disability index scale | 1-6 days
  A functional status scale ranging from 0% to 100% (0%= no activity limitation, 100% =complete activity limitation).
  Participants will be assessed immediately before and after treatment. Participants will be assessed 2 days per week with a minimum of 1 day between treatment days.

SECONDARY OUTCOMES:
Trends with use of perineural electrical dry needling with or without CGRP antagonist drugs. | following 4 weeks of treatment in the standard care plus perineural electrical dry needling arm.
  Because this is a small trial it is unlikely that we will be able to determine if migraine drugs significantly modify the effect perineural electrical dry needle treatment has on pain and the neck disability index. However we will look for any trends in interaction between perineural electrical dry needle treatment and migraine drugs using exploratory data analysis and box plot comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Joe Tepp, DPT, Principal Investigator — Ascension Healthcare
Locations (1):
- Ascension Rehabilitation Services, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04252391/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04252391/ICF_001.pdf